CLINICAL TRIAL: NCT04706000
Title: Investigation of Autophagy Markers in Endometrial Polyps
Brief Title: Autophagy Markers in Endometrial Polyps
Status: Completed | Type: Observational
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Burak Sezgin, Principal investigator M.D. Burak Sezgin, Muğla Sıtkı Koçman University
Other Study IDs: 03.09.20-08/01
Record Dates: First submitted 2021-01-08; First posted 2021-01-12 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Endometrial Polyp; Autophagy
Keywords: polyp; endometrium; beclin 1; LC3; p62
MeSH Terms: conditions — Polyps | interventions — Beclin-1

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: endometrial polyp
  Interventions: Genetic: Beclin 1 gene
- Control group: normal endometrium
  Interventions: Genetic: Beclin 1 gene

INTERVENTIONS:
Genetic: Beclin 1 gene — The determination of Beclin 1, LC3-II and p62 genes, which are evaluated by immunohistochemistry, at the protein level will be done by ELISA method in MSKU Medical Faculty Medical Biology Laboratory.
  Other Names: LC3-II gene; p62 gene

SUMMARY:
The aim of this research is to evaluate autophagy markers in patients with endometrial polyps

DETAILED DESCRIPTION:
Endometrial polyp are benign formations that are frequently encountered in gynecology practice and have malignant potential. It may be asymptomatic in the clinic or may present with abnormal uterine bleeding. Although its pathophysiology has not been clearly revealed, there are many studies in the literature about it. However, the autophagy pathway emerges as a subject that has never been evaluated. In this study, the investigators would like to prospectively evaluate Beclin 1, LC3A / B and p62 markers in the autophagy pathway in endometrial polyp tissue samples by immunohistochemistry and reveal their importance.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 35 years of age with a histopathologically confirmed diagnosis of endometrial polyp
* patients over the age of 35 whose histopathologically reported normal endometrial biopsy results.

Exclusion Criteria:

* Are under the age of 35,
* those with cognitive dysfunction,
* diagnosed with any type of cancer
* who are under treatment for cancer,
* diabetes mellitus,
* hypertension,
* endometriosis,
* adenomyosis,
* chronic endometritis,
* have an acute or chronic illness,
* patients who have smoked and used alcohol in the last 10 years

Min Age: 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — endometrial polyp
Study Population: Patients with histopathologically proven endometrial polyp and healthy controls
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2022-01-08 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
autophagy marker | through study completion, an average of 1 year
  Beclin 1 gene level
autophagy marker | through study completion, an average of 1 year
  LC3II gene level
autophagy marker | through study completion, an average of 1 year
  p62 gene level

CONTACTS AND LOCATIONS:
Overall Officials: Burak SEZGİN, MD, Principal Investigator — Muğla Sıtkı Koçman University
Locations (1):
- Mugla Sıtkı Kocman University Faculty of Medicine, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
When we conducted the study, we will plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Background] Zhang J. Teaching the basics of autophagy and mitophagy to redox biologists--mechanisms and experimental approaches. Redox Biol. 2015;4:242-59. doi: 10.1016/j.redox.2015.01.003. Epub 2015 Jan 13. PMID 25618581
- [Background] Zhan L, Yao S, Sun S, Su Q, Li J, Wei B. NLRC5 and autophagy combined as possible predictors in patients with endometriosis. Fertil Steril. 2018 Oct;110(5):949-956. doi: 10.1016/j.fertnstert.2018.06.028. PMID 30316442
- [Background] Xie Z, Klionsky DJ. Autophagosome formation: core machinery and adaptations. Nat Cell Biol. 2007 Oct;9(10):1102-9. doi: 10.1038/ncb1007-1102. PMID 17909521
- [Background] Wong M, Crnobrnja B, Liberale V, Dharmarajah K, Widschwendter M, Jurkovic D. The natural history of endometrial polyps. Hum Reprod. 2017 Feb;32(2):340-345. doi: 10.1093/humrep/dew307. Epub 2016 Dec 18. PMID 27994000
- [Result] Zhang L, Liu Y, Xu Y, Wu H, Wei Z, Cao Y. The expression of the autophagy gene beclin-1 mRNA and protein in ectopic and eutopic endometrium of patients with endometriosis. Int J Fertil Steril. 2015 Jan-Mar;8(4):429-36. doi: 10.22074/ijfs.2015.4183. Epub 2015 Feb 7. PMID 25780525